CLINICAL TRIAL: NCT03923985
Title: Clinical Trial to Evaluate the Effect of an Oral Probiotic (Food Supplement) Containing Lactobacillus Crispatus on the Vaginal Flora
Brief Title: Clinical Trial to Evaluate the Effect of an Oral Probiotic on the Vaginal Flora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Palacios (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SEID-Probiot
Record Dates: First submitted 2019-04-05; First posted 2019-04-23 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Vaginal Flora
Keywords: Vaginal Flora; Oral Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Arm (Active Comparator): 1 tablet / day of probiotic containing 10 Mld L. crispatus during two months
  Interventions: Dietary Supplement: Probiotic containing Lactobacillus Crispatus
- Control Arm (No Intervention): No treatment

INTERVENTIONS:
Dietary Supplement: Probiotic containing Lactobacillus Crispatus — 1 tablet / day of probiotic (275 mg of live probiotic lactic ferments: 10 Mld L. fermentum (SGL 10), 10 Mld L. gasseri, 10 Mld L. casei, 10 Mld L. acidophilus, 10 Mld L. crispatus) during 2 months.
  Arms: Active Arm

SUMMARY:
Clinical trial to evaluate the effect of a probiotic containing Lactobacillus Crispatus on the vaginal flora

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between 18 and 45 years old
* Women without current symptoms of vaginal infection
* Negative bacteriological and clinical examination

Exclusion Criteria:

* Women with vaginal infection
* Women with undiagnosed vaginal bleeding
* Patients with endometrial hyperplasia
* Suspicion of neoplasia or active neoplasia
* Women with intolerance, allergy or hypersensitivity to the components of the probiotic
* Women with immunosuppressive disorders or with HIV
* Women who are currently using probiotics by any route of administration
* Women who are using some treatment for vaginal sepsis
* Chronic decompensated noncommunicable diseases (diabetes mellitus, heart disease ...)
* Pregnant women or those with precocious menopause

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only Females
Enrollment: 40 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in the number of Lactobacillus Crispatus on the vaginal flora | Screening, month 2
  Analysis of vaginal lactobacilli.

SECONDARY OUTCOMES:
Changes in vaginal PH | Screening, month 2
  PH measurement

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Palacios, PhD, Principal Investigator — Instituto Palacios
Locations (1):
- Instituto Palacios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided